CLINICAL TRIAL: NCT06162117
Title: Validity and Reliability of the Two-Minute Step Test in Patients With Traumatic Meniscal Tear
Brief Title: Validity and Reliability of the Two-Minute Step Test in Traumatic Meniscal Tear
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRHmeniscus
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Meniscus Tear
Keywords: Exercise test; Meniscus; Physical fitness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic meniscus tear: Patients with traumatic meniscus tears will be enrolled in this study
  Interventions: Diagnostic Test: 2- Minute Step Test

INTERVENTIONS:
Diagnostic Test: 2- Minute Step Test — 2- Minute Step Test will be administered to patients with traumatic meniscus tear

SUMMARY:
This study is designed to explore the validity and reliability of the two-minute step test as an assessment method for functional capacity in patients diagnosed with traumatic meniscal tear. The objective is to determine the effectiveness of this test in accurately measuring the functional abilities of individuals with traumatic meniscus tears. By focusing on patients who have been diagnosed with such injuries and employing the two-minute step test, the study aims to provide valuable insights into the suitability of this evaluation tool for assessing functional capacity in this specific patient population. The findings of this research have the potential to contribute significantly to the clinical understanding and management of traumatic meniscal tears, offering clinicians a reliable and valid method for evaluating the functional capabilities of affected individuals.

DETAILED DESCRIPTION:
The study is planned as a cross-sectional clinical study. Fifty-five patients diagnosed with traumatic meniscal tear who apply to the Istanbul Physical Medicine and Rehabilitation Training and Research Hospital clinics will be included in the study. Patients must have a previous diagnosis of traumatic meniscal tear based on magnetic resonance imaging.

Sociodemographic data such as age, height, weight, body mass index, marital status, education level, and occupation will be recorded. The level of impairment in daily activities of patients with meniscal tear will be assessed using the Western Ontario Meniscus Evaluation Questionnaire. Pain intensity will be evaluated using the Visual Analog Scale, a linear scale of 10 cm. The Pain Catastrophizing Scale will be used to assess the patient's level of distress due to pain. The patient's confidence level in performing different activities due to pain will be evaluated using the Pain Self-Efficacy Questionnaire.

The patient's physical function will be assessed using the 2-Minute StepTest. This test, to be administered by the same evaluator, requires the patient to have rested for at least 30 minutes before starting, and there will be a minimum of 1 hour of rest between the tests conducted. Before starting the tests, the patient's blood pressure, oxygen saturation, and heart rate will be measured, and if results are outside the normal range, the test will not proceed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 50 who have previously been diagnosed with traumatic meniscal tear through magnetic resonance imaging will be included in the study

Exclusion Criteria:

* Patients under the age of 18 and over the age of 50
* Patients with accompanying knee osteoarthritis
* Degenerative meniscal tears
* Uncontrolled hypertension
* Decompensated cardiac failure
* Presence of systemic diseases affecting lower limb functions
* Presence of degenerative diseases affecting lower limb functions
* Peripheral artery disease causing vascular claudication
* Psychiatric illness
* Neuromuscular disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with traumatic meniscus tear
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Two-Minute Step Test | 0 day and 1th week
  During the administration of the Two-Minute Step Test, the midpoint between the anterior superior iliac spine and the patella of the patient is marked. The patient is then instructed to take steps in place as quickly as possible for a duration of two minutes. The knee should be lifted at least to the level of the marked point. The number of steps taken by the patient within the two-minute period is recorded.

SECONDARY OUTCOMES:
The Pain Self-Efficacy Questionnaire | 0 day
  The Pain Self-Efficacy Questionnaire comprises 10 items, with patients assigning confidence ratings on a scale from 0 points (indicating no confidence at all) to 6 points (indicating complete confidence). Total scores are computed by summing up the individual items, resulting in a score range from 0 points (indicating lower self-efficacy) to 60 points (indicating higher self-efficacy).
Pain Catastrophizing Scale | 0 day
  Individuals are required to express the extent to which they experience the thoughts and feelings mentioned above during pain using a scale of 0 (not at all) to 4 (all the time). The overall score ranges from 0 to 52, and it also provides three subscale scores evaluating rumination, magnification, and helplessness.
Western Ontario Meniscal Evaluation Tool | 0 day
  The Western Ontario Meniscal Evaluation Tool is a condition-specific instrument created for the assessment of Health-Related Quality of Life (HRQOL) in individuals with meniscal pathology. Comprising 16 items, it encompasses three domains. The physical symptom domain incorporates nine items, the combined domain covering sports, recreation, work, and lifestyle consists of four items, and the emotions domain includes three items.
  The best or least symptomatic score is 0, and the highest and most symptomatic score possible is 1,600.
Visual Analogue Scale | 0 day
  The Visual Analog Scale is a simple measurement tool consisting of a line with endpoints representing extreme points of a characteristic, such as "No Pain" to "Worst Pain Imaginable." Respondents mark a point on the line to indicate their perception or experience of the given characteristic. The distance from one endpoint to the marked point is then measured to quantify the subjective experience. It's commonly used to assess various subjective factors like pain, fatigue, or mood.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Physical Medicine and Rehabilitation Research and Training Hospital, Istanbul, Bahcelievler
  - Beylikdüzü State Hospital, Istanbul, Beylikdüzü

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliveros MJ, Seron P, Roman C, Galvez M, Navarro R, Latin G, Marileo T, Molina JP, Sepulveda P, Marzuca-Nassr GN, Munoz S. Two-Minute Step Test as a Complement to Six-Minute Walk Test in Subjects With Treated Coronary Artery Disease. Front Cardiovasc Med. 2022 May 9;9:848589. doi: 10.3389/fcvm.2022.848589. eCollection 2022. PMID 35615563
- [Result] de Jesus SFC, Bassi-Dibai D, Pontes-Silva A, da Silva de Araujo A, de Freitas Faria Silva S, Veneroso CE, de Paula Gomes CAF, Dibai-Filho AV. Construct validity and reliability of the 2-Minute Step Test (2MST) in individuals with low back pain. BMC Musculoskelet Disord. 2022 Dec 5;23(1):1062. doi: 10.1186/s12891-022-06050-w. PMID 36471309
- [Result] de Morais Almeida TF, Dibai-Filho AV, de Freitas Thomaz F, Lima EAA, Cabido CET. Construct validity and reliability of the 2-minute step test in patients with knee osteoarthritis. BMC Musculoskelet Disord. 2022 Feb 17;23(1):159. doi: 10.1186/s12891-022-05114-1. PMID 35177048